CLINICAL TRIAL: NCT02681796
Title: Epidural Analgesia Use in Pancreatic Resections
Acronym: E-PRO I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201506125
Record Dates: First submitted 2016-02-10; First posted 2016-02-12 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Cancer of Pancreas; Cancer of the Pancreas; Pancreas Cancer; Pancreas Neoplasms; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study: Bupivacaine Epidural + standard of care pain regimen (Experimental): -The study group will receive a T6 to T8 level epidural catheter in addition to the standardized pain regimen. Epidurals used in this study will contain a 0.125% bupivacaine-only infusion
  Interventions: Drug: Bupivacaine
- Control: Standard of care pain regimen (No Intervention): -The control group will receive a standardized pain regimen including an opioid patient controlled analgesia (PCA), IV acetaminophen, and IV ketorolac per surgeon's preference

INTERVENTIONS:
Drug: Bupivacaine
  Arms: Study: Bupivacaine Epidural + standard of care pain regimen

SUMMARY:
The rationale for this study is to investigate the benefits of epidural analgesia in pancreatic resections in a prospective, single blind, randomized control trial. This study will evaluate both short and long-term outcomes related to epidural analgesia, providing a longitudinal and comprehensive perspective to the advantages and disadvantages of this technique. The investigators hypothesize that the use of epidural analgesia reduces a patient's consumption of morphine or morphine-equivalent in the post-operative period following pancreatic resections.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing pancreatic resection.
* Age ≥18 years old.
* Able to understand and sign an Institutional Review Board (IRB)-approved informed consent form.

Exclusion Criteria:

* Indication for operative intervention being chronic pancreatitis.
* Currently on warfarin with an INR≥1.4 or clopidogrel that cannot be discontinued 7 days prior to surgery;
* Most recent INR prior to surgery >1.4
* Most recent platelet count prior to surgery <70,000/mcl
* Chronic opioid use as defined by use of more than 20mg oxycodone, or equivalent, daily.
* History of pre-existing neuropathic pain conditions.
* Not giving consent for study participation.
* Known medical history of significant psychiatric or cognitive impairment
* History of HIV, Hepatitis B, and/or Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Total consumption of morphine or morphine-equivalent in patients undergoing pancreatic resections in the control group compared with the study group | First 72 hours after surgery
  -Will be assessed every 24 hours

SECONDARY OUTCOMES:
Effect of epidural analgesia during the initial post-operative period as measured by total intraoperative fluid volume | During surgery
Benefit of epidural analgesia as measured by the reduction of persistent post-surgical pain (PPSP) after the operation | Up to 6 weeks post-surgery
  -Quantitative sensory testing will be performed on the abdomen in close proximity to the surgical incision
Benefit of epidural analgesia as measured by time to tumor recurrence | Up to 2 years post surgery
Benefit of epidural analgesia as measured by disease-free survival | Up to 2 years post surgery
Benefit of epidural analgesia as measured by overall survival | Up to 2 years post surgery
Rate of delirium in the control group compared with the study group | First 72 hours after surgery
  * Assessed for delirium using the 3D-CAM instrument
  * Postoperative delirium assessments will be performed when patients can be around sufficiently in order to be assessed for delirium using the Richmond-Agitation-Sedation Scale.
  * Will be assessed for delirium once daily in the afternoon/evening
Effect of epidural analgesia during the initial post-operative period as measured by total post-operative fluid volume | Up to 72 hours post surgery
Effect of epidural analgesia during the initial post-operative period as measured by volume of fluid boluses | Up to 72 hours post surgery
Effect of epidural analgesia during the initial post-operative period as measured by amount of antiemetic doses | Up to 72 hours post surgery
Effect of epidural analgesia during the initial post-operative period as measured by return of bowel function by time to first flatus | Up to 72 hours post surgery
Effect of epidural analgesia during the initial post-operative period as measured by first bowel movement | Up to 72 hours post surgery
Effect of epidural analgesia during the initial post-operative period as measured by length of hospital stay | Up to 2 weeks post surgery
Effect of epidural analgesia during the initial post-operative period as measured by incidence of deep venous thromboembolism/pulmonary embolism | Up to 72 hours post surgery
Effect of epidural analgesia during the initial post-operative period as measured by relative ratios of blood level inflammatory markers | Up to 6 weeks post-surgery
  -Specifically interleukin-1-beta (IL-1B), interleukin-6 (IL-6), tumor necrosis factor-alpha (TNF-a), and interleukin 10 (IL-10) biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bottros, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pak LM, Haroutounian S, Hawkins WG, Worley L, Kurtz M, Frey K, Karanikolas M, Swarm RA, Bottros MM. Epidurals in Pancreatic Resection Outcomes (E-PRO) study: protocol for a randomised controlled trial. BMJ Open. 2018 Jan 26;8(1):e018787. doi: 10.1136/bmjopen-2017-018787. PMID 29374667
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu